CLINICAL TRIAL: NCT01850251
Title: Randomized Controlled, Pilot Study to Assess the Effect of a High Protein and Calorie Nutritional Supplementation Enriched Hydroxymethylbutyrate and Vitamin D on Muscle Strength and Function in Patients With Hip Fracture.
Brief Title: Effects of a Supplement Enriched in Hydroxymethylbutyrate and Vitamin D on Muscle Strength in Hip Fracture
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruiting problems.
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Pere Leyes, Specialist, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ORTOHMB-13
Record Dates: First submitted 2013-05-03; First posted 2013-05-09 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Hip Fractures
Keywords: Hip fractures; Ageing; Sarcopenia; Function
MeSH Terms: conditions — Hip Fractures; Sarcopenia | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplement with HMB and vitamin D (Experimental): Oral administration of 440 mL (2 bottles) of nutritional supplement with HMB and vitamin D each day during 8 weeks.
  Interventions: Dietary Supplement: Supplement with HMB and vitamin D
- Standard nutritional supplement (Active Comparator): Oral administration of 440 mL (2 bottles) of standard nutritional supplement each day during 8 weeks.
  Interventions: Dietary Supplement: Standard nutritional supplement

INTERVENTIONS:
Dietary Supplement: Supplement with HMB and vitamin D — High protein, high calorie nutritional supplement enriched with hydroxymethylbutyrate and vitamin D.
  Other Names: Ensure Plus Advance
  Arms: Supplement with HMB and vitamin D
Dietary Supplement: Standard nutritional supplement — High protein, high calorie nutritional supplement.
  Other Names: Ensure Plus High Protein
  Arms: Standard nutritional supplement

SUMMARY:
The purpose of this study is to determine whether a nutritional supplement high in protein and energy, and enriched with hydroxymethylbutyrate (HMB) and vitamin D is more effective than a standard nutritional supplement high in protein and energy in improving muscle strength in elderly patients with hip fracture.

DETAILED DESCRIPTION:
Hip fractures are the cause of substantial morbidity and mortality in elderly people. Nine months after hip fracture, patients still have a poorer quality of life compared to control subjects matched for age and sex.

After a hip fracture, many patients fail to return to their homes and their previous state of mobility. Acute hospital costs generated by this condition are substantial, although the costs in rehabilitation and special care in long-term community are even greater.

Patients with hip fracture are most likely to be frail elderly, and they are usually malnourished when the fracture occurs. Moreover, physiological aging is accompanied by functional losses and changes in the various organs and systems, including the musculoskeletal system, in which there is a progressive reduction of muscle mass, called sarcopenia. Approximately 30% of muscle mass is lost between the fifth and eighth decades of life and the percentage of muscle loss can reach 15% per decade after 70 years of age. Having established a correlation between the loss of muscle mass and loss of strength, sarcopenia has been associated with a risk of functional disability twice in men and thrice in women.

Hydroxymethylbutyrate (HMB) is a leucine metabolite produced in small quantities (0.3-0.4 g/d). Leucine effects on muscle metabolism appear to be due, in part, to HMB. In vitro experiments have observed that HMB attenuates proteolysis processes through the inhibition of various catabolic pathways and could stimulate protein synthesis. There are some evidences that administration of HMB in the elderly results in increases in muscle strength and functionality enhancements, compared to a control group.

In elderly people, low levels of vitamin D have been associated, among others, to decreased muscle strength, falls and fractures. The elderly have an increased risk of developing vitamin D deficiency due to less sun exposure, a decrease in the absorption and changes in the metabolism of this vitamin. Because muscle weakness is a clinical feature of vitamin D deficiency, it has been postulated that its deficiency could precipitate and increase muscle weakness and functional decline in older people.

Therefore, the study raises the possibility that an intervention consisting of a high protein, high calorie oral nutritional supplement enriched with HMB and vitamin D is more effective than a standard high protein, high calorie oral nutritional supplement in improving muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years of age after hip fracture surgery.
* Ability to walk before fracture.

Exclusion Criteria:

* Chronic renal failure, defined as a glomerular filtration rate less than 60 mL/min/1.73 m2, or serum creatinine of 0.9 mg/dL in women or 1.2 mg/dL in men.
* Following a diet with protein restriction.
* Need for enteral or parenteral nutrition.
* Need for medication with orexigenic or anabolic effect, or long-term corticosteroids.
* Active neoplastic disease.
* Cognitive impairment or major psychiatric disorder.
* Lack of signed informed consent.
* Any patient with inability to comply with treatment or not appropriate according to the investigator.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in bilateral knee extension test as a measure of isometric muscle strength. | Baseline and 8 weeks
  Changes from baseline in the knee extension test at 8 weeks will be conducted using a dynamometer.

SECONDARY OUTCOMES:
Change in the Timed Up & Go test as a measure of function. | Baseline and 8 weeks
  Changes from baseline in the Timed Up & Go functional test at 8 weeks.

OTHER OUTCOMES:
Quality of life | Baseline and 8 weeks
  Change from baseline in quality of life at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Forga, MD, Principal Investigator — Hospital Clinic of Barcelona; Joan Trabal, RD, MS, Study Chair — Hospital Clinic of Barcelona; Pere Leyes, MD, Study Chair — Hospital Clinic of Barcelona; Salvi Prat, MD, PhD, Study Chair — Hospital Clinic of Barcelona; Margarita Navarro, MD, Study Chair — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Catalonia, Spain

REFERENCES:
- [Background] Fuller JC Jr, Baier S, Flakoll P, Nissen SL, Abumrad NN, Rathmacher JA. Vitamin D status affects strength gains in older adults supplemented with a combination of beta-hydroxy-beta-methylbutyrate, arginine, and lysine: a cohort study. JPEN J Parenter Enteral Nutr. 2011 Nov;35(6):757-62. doi: 10.1177/0148607111413903. Epub 2011 Aug 1. PMID 21807930